CLINICAL TRIAL: NCT05566483
Title: Physiological Underpinnings of Post-Acute Sequelae of SARS CoV-2 ("Long COVID") and Impact of Cardiopulmonary Rehabilitation on Quality-of-Life and Functional Capacity
Brief Title: Physiology of Long COVID-19 and the Impact of Cardiopulmonary Rehabilitation on Quality-of-Life and Functional Capacity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-1093
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Post-acute Sequelae of SARS-CoV-2 Infection
Keywords: Cardiopulmonary Rehabilitation; Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — exercise protocol
  Arms: Exercise

SUMMARY:
The primary objectives of this study are to determine whether exercise training is an effective strategy for treatment of Long COVID and characterize the cardiorespiratory and autonomic physiology in these patients to precisely characterize mechanisms contributing to this syndrome.

DETAILED DESCRIPTION:
Abnormalities observed among Long COVID patients are consistent with cardiac deconditioning. The Long COVID syndrome has been attributed to dysautonomia and/or postural orthostatic tachycardia syndrome (POTS) based largely on anecdotal experience and observations of positional tachycardia among affected individuals. However, it has been emphasized that data are clearly lacking to implicate dysautonomia alone as the cause of Long COVID. Alternatively, cardiac deconditioning leads to a constellation of symptoms, including exercise intolerance, brain fog/cognitive impairments, tachycardia and orthostatic intolerance, all of which are reported among reported among patients with Long COVID. Multiple studies have demonstrated that cardiac deconditioning may occur with as little as 20 hours of bedrest. Exercise training improves cardiorespiratory performance among patients suffering from cardiac deconditioning. Exercise training improves HR regulation and cardiovascular function during submaximal and peak exercise, and improves overall exercise capacity particularly among individuals with cardiac deconditioning following bedrest (e.g. Dallas bedrest studies) and among individuals with postural orthostatic tachycardia syndrome. Our preliminary data demonstrate a significant improvement/resolution in Long-COVID symptoms following a twelve-week exercise training program in a community setting. During the height of the COVID pandemic, the investigators developed an exercise protocol that has been used in the clinical setting to assist with management of patients suffering from Long COVID. This protocol involves recumbent/semi-recumbent exercise - specifically, rowing or cycling on a recumbent ergometer.

This proposal involves a clinical trial involving a two-aim initiative whereby participants with Long COVID will be randomized to a 12-week period of exercise training v. usual care ("controls") with baseline and follow-up assessments in order to: 1) Determine whether exercise training is an effective treatment strategy for management of Long COVID (Aim 1); and 2) Characterize cardiovascular/autonomic physiology among patients with Long COVID (Aim 2). In a third aim, healthy individuals will undergo a hemodynamic assessment afterbefore and after 24 hours of bedrest. The hemodynamic assessment will be identical to participants with Long COVID.

There will be a baseline assessment (Visit1) for all participants. After the baseline assessment, participants will be randomized in a 1:1 fashion to either undergo an exercise training program (exercise group) or usual care (control group) with no intervention. After completion of the exercise training program, the exercise group will return for a follow-up assessment (Visit2) that will be identical to the baseline (Visit 1) assessment. Participants in the control group will return for a follow-up (Visit 2) assessment, after which time they will crossover to complete the exercise training program. After completion of the exercise training program, these participants will return for a follow-up assessment (Visit 3). So, participants in the exercise group will complete two visits; participants in the control group will complete three visits.

Each assessment (Visits 1,2 and 3) is identical and includes a baseline resting assessment, watching heart rate and blood pressure while laying flat, as well as a tilt table test, a 10-minute stand, and an exercise test. Participants also complete a questionnaire asking about quality-of-life. The visit lasts about 2-2.5 hours.

The exercise training program is about twelve weeks long. Participants are provided exercise equipment at home, to complete the program. The program involves recumbent exercise (e.g. rowing machine, or recumbent cycling) and starts off with low duration, low intensity exercise, and gradually increases in duration and intensity over time.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with documented history of COVID-19 infection and symptoms consistent with Long COVID lasting >12 weeks after diagnosis.

Exclusion Criteria:

* History of cardiovascular/pulmonary disease prior to infection
* COVID-related myocardial injury such as evidence of myocarditis
* Deep vein thrombosis/pulmonary embolism following COVID-19 infection
* Exercise intolerance resulting from conditions that are not related to cardiorespiratory or autonomic factors (e.g. osteoarthritis or other musculoskeletal diseases);
* Dependency of supplemental oxygen following COVID infection due to cardiovascular and/or pulmonary complications following acute COVID infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Characterizing the impact of exercise training (cardiac rehabilitation) on functional capacity among patients with Long COVID | 12 weeks
  functional capacity as determined by VO2max
Characterizing the impact of exercise training (cardiac rehabilitation) on HRqOL among patients with Long COVID | 12 weeks
  Health-related quality of life (HRqOL) from SF-36 form; all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.

SECONDARY OUTCOMES:
orthostatic challenge | 12 weeks
  Heart rate during orthostatic challenge

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larsen NW, Stiles LE, Miglis MG. Preparing for the long-haul: Autonomic complications of COVID-19. Auton Neurosci. 2021 Nov;235:102841. doi: 10.1016/j.autneu.2021.102841. Epub 2021 Jul 3. PMID 34265539
- [Background] Writing Committee; Gluckman TJ, Bhave NM, Allen LA, Chung EH, Spatz ES, Ammirati E, Baggish AL, Bozkurt B, Cornwell WK 3rd, Harmon KG, Kim JH, Lala A, Levine BD, Martinez MW, Onuma O, Phelan D, Puntmann VO, Rajpal S, Taub PR, Verma AK. 2022 ACC Expert Consensus Decision Pathway on Cardiovascular Sequelae of COVID-19 in Adults: Myocarditis and Other Myocardial Involvement, Post-Acute Sequelae of SARS-CoV-2 Infection, and Return to Play: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2022 May 3;79(17):1717-1756. doi: 10.1016/j.jacc.2022.02.003. Epub 2022 Mar 16. No abstract available. PMID 35307156
- [Background] Mitchell JH, Levine BD, McGuire DK. The Dallas Bed Rest and Training Study: Revisited After 50 Years. Circulation. 2019 Oct 15;140(16):1293-1295. doi: 10.1161/CIRCULATIONAHA.119.041046. Epub 2019 Oct 14. No abstract available. PMID 31609661
- [Background] Saltin B, Blomqvist G, Mitchell JH, Johnson RL Jr, Wildenthal K, Chapman CB. Response to exercise after bed rest and after training. Circulation. 1968 Nov;38(5 Suppl):VII1-78. No abstract available. PMID 5696236
- [Background] Mancini DM, Brunjes DL, Lala A, Trivieri MG, Contreras JP, Natelson BH. Use of Cardiopulmonary Stress Testing for Patients With Unexplained Dyspnea Post-Coronavirus Disease. JACC Heart Fail. 2021 Dec;9(12):927-937. doi: 10.1016/j.jchf.2021.10.002. PMID 34857177